CLINICAL TRIAL: NCT07174557
Title: Beyond the Clinic: Enhancing Depression Surveillance With a Digital Biomarker
Brief Title: Remote Evaluation and Alerting for Collaborative Health (REACH) in Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nicholas C. Jacobson, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00033020; 5UM1TR004772-02 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Smartphone monitoring; Risk detection; Collaborative care
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: Sensing System Calibration (N = 120) (Experimental): We expect that participants will be in this research study for six months. Participants will be asked to download an app on their smartphone. This app will collect data from the phone's sensors. Participants will also be asked to answer some questions about their mood each month.
  Interventions: Other: MoodTriggers Application
- Phase 2: Early warning system (n = 100) (Active Comparator): This study is randomized which means that in order to learn about the effect of the Smartphone App, half the people in this study will use it, and the other half will not. If participants decide to enroll into this research study, they may be assigned by chance to download a Smartphone App. This App will collect data from the phone's sensors. Participants will also be asked to complete questionnaires about their mood each month.
  Interventions: Other: MoodTriggers Application
- Phase 2: Usual Care (n = 100) (No Intervention): This study is randomized which means that in order to learn about the effect of the Smartphone App, half the people in this study will use it, and the other half will not. If participants decide to enroll into this research study, they may be assigned by chance to have usual care. Participants will be asked to complete questionnaires about their mood each month.

INTERVENTIONS:
Other: MoodTriggers Application — The Mood Triggers application, developed by Dr. Jacobson, will be used for collecting smartphone sensor data. This HIPAA-compliant app has been incorporated into various projects at Dartmouth, Stanford, and MGH/Harvard, with development supported by NIDA, NIMHD, NCI, and the Department of Veterans Affairs. The Mood Triggers app will capture a wide range of metrics, including psychomotor agitation, sleep disturbances, low behavioral activation, social contact, exposure to natural light, heart rate, heart rate variability, and screen time. The app also tracks the patient's screen time and app usage data. The Mood Triggers App will be installed on the smartphones at time of informed consent for all 120 patients enrolled in Phase 1 and for 100 clinical trial participants randomized to the "early warning system" (intervention arm) in Phase 2. Data will be collected from the Mood Triggers App starting on day of discharge from care and for 6 months post-discharge date.
  Arms: Phase 1: Sensing System Calibration (N = 120); Phase 2: Early warning system (n = 100)

SUMMARY:
Researchers hope to see if the data smartphones collect continuously can be used to predict if patient's depression symptoms will return. They will do this by collecting data from patient's smartphones and comparing it to their depression symptoms. If this method is successful, researchers could develop a smartphone application to help healthcare providers better monitor patient's depression and intervene earlier if symptoms return.

DETAILED DESCRIPTION:
Study phase 1: The investigators expect that participants will be in this research study for six months. Participants will be asked to download an app on their smartphone. This app will collect data from the phone's sensors. Participants will also be asked to answer some questions about their mood each month.

Study phase 2: This phase of the study is randomized which means that in order to learn about the effect of the Smartphone App, half the people in this study will use it, and the other half will not. If participants decide to enroll into this research study, they will be assigned by chance to one of the following groups:

Group A: Participants will be asked to download a Smartphone App. This App will collect data from the phone's sensors.

Group B: Participants will have usual care. Both Groups: Participants will be asked to complete questionnaires about their mood each month.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Treated for depression within Dartmouth Health collaborative care model (CoCM) sites who are discharged from CoCM without depression (PHQ-9 < 10)
* Have access to and ability to use a smartphone (Android version ≥ 6 or iOS version ≥ 11).

Exclusion Criteria:

* Identified as high risk due to active suicidality, psychosis, or bipolar disorder - Discharged from CoCM with ongoing depressive symptoms (PhQ-9 > 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Monthly depression relapse | discharge, 6-months post-discharge
  The 9-item Patient Health Questionnaire (PHQ-9), a validated self-reported depression questionnaire, will be used to detect monthly depression recurrence based on past-month MoodTriggers application data. The PHQ-9 scores range from 0-27, with higher scores reflecting higher depression symptom levels. The PHQ-9 will be used to detect monthly recurrence of Major Depressive Disorder (MDD; PHQ-9 scores ≥ 10) during Phase 1 in all 120 participants. For the randomized clinical trial in Phase 2, we will capture the PHQ-9 monthly in both arms (MoodTriggers app vs. no app) for 6-months following discharge.

SECONDARY OUTCOMES:
Perceived benefits and barriers of depression monitoring using passive sensing data collected from mobile phones | 0-6 months post-discharge
  A subgroup of individuals from Phase 1 will be invited and verbally consented to participate in semi-structured interviews to provide their experiences with the study's digital biomarker "early warning" system. The purpose of this interview is to identify perceived benefits and barriers of depression monitoring using passive sensing data collection from your mobile phone. The information gathered will be used to evaluate the effectiveness of the Mood Trigger app in predicting symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Jacobson, PhD, Principal Investigator — Dartmouth College
Locations (2):
- United States (2):
  - Dartmouth College, Hanover, New Hampshire
  - Dartmouth-Hitchcock Clinics, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No